CLINICAL TRIAL: NCT01439048
Title: Study of Environmental Toxicants and Inflammatory Markers in Prematurity and Diseases of Prematurity
Brief Title: Placental and Cord Blood Markers Associated With Premature Birth and Disorders of Premature Birth in Newborn Infants
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Venkatesh Sampath, Staff Physician, Medical College of Wisconsin
Other Study IDs: CHW 09/102, GC 900
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Premature Birth
Keywords: Placenta; Cord Blood; PAH; Environmental Markers; Toll-Like Receptors
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, placenta
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Term infants: Infants born at greater than 37 weeks gestation
- Preterm Infants: Infants born at less than 37 weeks gestation

SUMMARY:
The purpose of this study is to determine if changes in specific gene products in the placenta or cord/infant blood affect a baby's birth weight, increase the risk of premature birth, or increase the risk of developing diseases of prematurity. We would also like to characterize whether placental epigenetic changes or placental markers of environmental exposures are associated with premature birth.

DETAILED DESCRIPTION:
Prematurity, diseases of prematurity and growth-disorders of newborn infants contribute significantly to morbidity and mortality seen in newborn infants [1,2,3]. One out of eight newborn infants in the USA is born premature (gestational age less than 37 completed weeks). In 2004, of the 27,860 infants dying within the first year of life, greater than 16,000 were born premature [2]. Moreover, premature infants who survive the neonatal period are at increased risk of cerebral palsy, developmental delays, growth impairment and long-term respiratory disability [3-5]. Additionally, fetal growth restriction and fetal growth excess results in infants being delivered as small for gestational age infants or large for gestational age infants, respectively. Infants born with such growth-disorders are at increased risk of perinatal morbidity and mortality and as adults are at significant risk of obesity, type II diabetes and heart disease [6,7].

While the etiology of preterm birth and growth-disorders can be ascribed to maternal conditions, chromosomal defects or specific maternal environmental exposures in some newborn infants, for a majority the etiology remains unknown [8,9]. There is increasing evidence pointing to the role of genetic susceptibility factors in the causation of prematurity and growth-disorders of the newborn infant [8, 10-12]. Further, epigenetic changes in growth regulating or inflammatory genes in the placenta can program the fetus for premature birth, growth-disorders and other diseases in the postnatal period.

The overall objective of this application is four-fold.

1. To determine whether altered placental or fetal expression of imprinted genes is associated with disorders of growth, prematurity or other postnatal diseases in newborn infants.
2. To determine whether altered placental expression of genes that regulate the innate immune response is associated with premature birth or other postnatal diseases in newborn infants.
3. To determine whether placental markers of environmental exposure (such as Polycyclic Aromatic Hydrocarbons or PAH) or epigenetic changes in placental inflammatory genes or growth genes are associated with prematurity or postnatal diseases in newborn infants.
4. To determine whether cord blood immune responses and markers of immune-cell function are different between preterm and term infants and are associated with postnatal diseases in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* all infants born alive

Exclusion Criteria:

* infants who are born with no signs of life

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who are born both premature (less than 37 weeks gestation) and full term infants (greater than 37 weeks gestation).
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Comparisons of placental gene expression and cord blood immune markers | through hospital discharge
  Placental gene expression and cord-blood immune markers/function will be compared between 50 term infants and 150 preterm infants. Further, among preterm infants it will be determined whether certain patterns of gene expression and immune marker distribution are associated with specific diseases/condition and growth outcomes. Similarly, epigenetic changes in the immune genes and markers of environmental exposure will be compared between preterm infants and term infants. Associations between environment exposures and epigenetic changes and diseases of prematurity will also be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Sampath, MBBS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Wauwatosa, Wisconsin, United States

REFERENCES:
- [Background] Guyer B, Martin JA, MacDorman MF, Anderson RN, Strobino DM. Annual summary of vital statistics--1996. Pediatrics. 1997 Dec;100(6):905-18. doi: 10.1542/peds.100.6.905. PMID 9374556
- [Background] Mathews TJ, MacDorman MF. Infant mortality statistics from the 2003 period linked birth/infant death data set. Natl Vital Stat Rep. 2006 May 3;54(16):1-29. PMID 16711376
- [Background] Stoll BJ, Hansen N. Infections in VLBW infants: studies from the NICHD Neonatal Research Network. Semin Perinatol. 2003 Aug;27(4):293-301. doi: 10.1016/s0146-0005(03)00046-6. PMID 14510320
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Background] Chakraborty S, Joseph DV, Bankart MJ, Petersen SA, Wailoo MP. Fetal growth restriction: relation to growth and obesity at the age of 9 years. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F479-83. doi: 10.1136/adc.2006.109728. Epub 2007 Feb 14. PMID 17301112
- [Background] Valsamakis G, Kanaka-Gantenbein C, Malamitsi-Puchner A, Mastorakos G. Causes of intrauterine growth restriction and the postnatal development of the metabolic syndrome. Ann N Y Acad Sci. 2006 Dec;1092:138-47. doi: 10.1196/annals.1365.012. PMID 17308140
- [Background] Adams KM, Eschenbach DA. The genetic contribution towards preterm delivery. Semin Fetal Neonatal Med. 2004 Dec;9(6):445-52. doi: 10.1016/j.siny.2004.04.001. PMID 15691782
- [Background] Kramer MS. Intrauterine growth and gestational duration determinants. Pediatrics. 1987 Oct;80(4):502-11. PMID 3658568
- [Background] Hao K, Wang X, Niu T, Xu X, Li A, Chang W, Wang L, Li G, Laird N, Xu X. A candidate gene association study on preterm delivery: application of high-throughput genotyping technology and advanced statistical methods. Hum Mol Genet. 2004 Apr 1;13(7):683-91. doi: 10.1093/hmg/ddh091. Epub 2004 Feb 19. PMID 14976157
- [Background] Clausson B, Lichtenstein P, Cnattingius S. Genetic influence on birthweight and gestational length determined by studies in offspring of twins. BJOG. 2000 Mar;107(3):375-81. doi: 10.1111/j.1471-0528.2000.tb13234.x. PMID 10740335
- [Background] Treloar SA, Macones GA, Mitchell LE, Martin NG. Genetic influences on premature parturition in an Australian twin sample. Twin Res. 2000 Jun;3(2):80-2. doi: 10.1375/136905200320565526. PMID 10918619